CLINICAL TRIAL: NCT05303532
Title: ROSY-D: Roll Over StudY for Patients Who Have Completed a Previous Oncology Study With Durvalumab and Are Judged by the Investigator to Clinically Benefit From Continued Treatment
Brief Title: Roll Over StudY for Patients Who Have Completed a Previous Oncology Study With Durvalumab
Acronym: ROSY-D
Status: Enrolling by invitation | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: D4191C00137; 2021-003031-29 (EudraCT Number)
Record Dates: First submitted 2022-02-04; First posted 2022-03-31 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Cancer
Keywords: Cancer; Oncology; Clinically Benefit; Roll Over StudY; Durvalumab
MeSH Terms: conditions — Neoplasms | interventions — durvalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Durvalumab (Experimental): Participants will receive durvalumab.
  Interventions: Drug: Durvalumab

INTERVENTIONS:
Drug: Durvalumab — Fixed dose of 1500 mg via IV infusion upon enrollment visit and every 4 weeks thereafter.

SUMMARY:
The rationale of the ROSY-D study is to continue to provide study treatment for patients who have participated in a parent study with Durvalumab and who are continuing to derive clinical benefit from treatment at the end of such studies, as judged by the Investigator.

DETAILED DESCRIPTION:
ROSY-D is an open label, non-randomised, multicentre, international trial for patients who have completed a parent study using durvalumab and who are deriving clinical benefit from continued treatment as judged by the Investigator. Patients will be rolled-over from the parent study and will continue the study indefinitely, until they meet one of the treatment discontinuation criteria.

ELIGIBILITY:
Inclusion Criteria:

The Core Protocol inclusion criteria are:

* Provision of signed and dated, written Informed Consent Form (ICF).
* Patient is currently deriving clinical benefit, as judged by the investigator, from continued treatment in an AstraZeneca parent study using an AstraZeneca compound that has met its endpoints, or has otherwise stopped, or the patient has reached maximum treatment duration allowed in the parent study's protocol.
* Patient can receive durvalumab as a fixed dose of 1500 mg quarterly 4 weeks at study entry.

There are no additional inclusion criteria for the ROSY-D sub-study.

Exclusion Criteria:

The Core Protocol exclusion criteria are.

* Ongoing, unresolved, Grade 3 or above toxicity requiring interruption of treatment at the time of the termination of the parent study.
* Currently receiving treatment with any prohibited medication(s).
* Concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study.
* Permanent discontinuation from the parent study due to toxicity or disease progression (increase in the severity of the disease under study and/or increases in the symptoms of a patient's condition attributable to the disease, as assessed and documented by the Investigator. Physician-defined progression can be radiological [example: Response Evaluation Criteria in Solid Tumours] progression or clinical progression).
* Local access to commercially-available drug at no cost to the patient as permitted by local/country regulation.

The additional exclusion criteria for the ROSY-D sub-study are:

* Active infection including Coronavirus disease 2019 (Polymerase chain reaction confirmed and/or clinically suspected), tuberculosis, hepatitis B (known positive Hepatitis B virus (HBV) surface antigen result), hepatitis C, or Human immunodeficiency virus (HIV) (positive HIV 1/2 antibodies).
* Male or female patients of reproductive potential who are not willing to employ effective birth control from study inclusion up to 90 days after the last dose of durvalumab monotherapy.
* Ongoing, unresolved, Grade 2 toxicity with an inability to reduce corticosteroid to a dose of ≤ 10 mg of prednisone per day (or equivalent) within 12 weeks after last dose of study treatment/study regimen, per Toxicity Dose Modification and TMGs for Immune- mediated, Infusion-related, and Non-Immune-mediated Reactions Guidelines of the parent study.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Estimated)
Dates: Start 2022-04-19 (Actual); Primary Completion 2026-01-07 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with serious adverse events as assessed by Common Terminology Criteria for Adverse Events (CTCAE) v5.0 | From baseline up to follow up at 90 days after the last dose of study drug.
  To monitor safety and tolerability of continuous study treatment to patients who continue to benefit at the end of the clinical trial by measuring the primary outcome of Serious Adverse Events (SAEs).

CONTACTS AND LOCATIONS:
Locations (113):
- United States (3):
  - Research Site, Newport Beach, California
  - Research Site, Denver, Colorado
  - Research Site, Memphis, Tennessee
- Research Site, Rosario, Argentina
- Australia (2):
  - Research Site, Box Hill
  - Research Site, Melbourne
- Research Site, Charleroi, Belgium
- Brazil (2):
  - Research Site, Barretos
  - Research Site, São José do Rio Preto
- Research Site, Sofia, Bulgaria
- Canada (3):
  - Research Site, Kingston, Ontario
  - Research Site, Newmarket, Ontario
  - Research Site, Toronto, Ontario
- China (9):
  - Research Site, Beijing
  - Research Site, Changsha
  - Research Site, Hangzhou
  - Research Site, Nanjing
  - Research Site, Shanghai
  - Research Site, Shenyang
  - Research Site, Wenzhou
  - Research Site, Xi'an
  - Research Site, Xiamen
- Research Site, Olomouc, Czechia
- France (14):
  - Research Site, Besançon
  - Research Site, Bordeaux
  - Research Site, Brest
  - Research Site, Dijon
  - Research Site, Lyon
  - Research Site, Marseille
  - Research Site, Montpellier
  - Research Site, Rennes
  - Research Site, Rouen
  - Research Site, Saint-Herblain
  - Research Site, Strasbourg
  - Research Site, Toulouse
  - Research Site, Tours
  - Research Site, Villejuif
- Germany (3):
  - Research Site, Gütersloh
  - Research Site, Münster
  - Research Site, Oldenburg
- Research Site, Athens, Greece
- Hungary (3):
  - Research Site, Budapest
  - Research Site, Győr
  - Research Site, Székesfehérvár
- Research Site, Chennai, India
- Italy (9):
  - Research Site, Arezzo
  - Research Site, Bari
  - Research Site, Catania
  - Research Site, Meldola
  - Research Site, Milan
  - Research Site, Modena
  - Research Site, Padua
  - Research Site, Pisa
  - Research Site, Roma
- Japan (8):
  - Research Site, Bunkyō City
  - Research Site, Fukuoka
  - Research Site, Kanazawa
  - Research Site, Kōtoku
  - Research Site, Nagoya
  - Research Site, Okayama
  - Research Site, Saga
  - Research Site, Sunto-gun
- Research Site, Kuching, Malaysia
- Mexico (3):
  - Research Site, Aguascalientes
  - Research Site, Mexico City
  - Research Site, Mérida
- Research Site, Quezon City, Philippines
- Poland (7):
  - Research Site, Bialystok
  - Research Site, Bydgoszcz
  - Research Site, Elblag
  - Research Site, Lodz
  - Research Site, Olsztyn
  - Research Site, Szczecin
  - Research Site, Warsaw
- Research Site, Suceava, Romania
- Russia (5):
  - Research Site, Moscow
  - Research Site, Nizhny Novgorod
  - Research Site, Novosibirsk
  - Research Site, Omsk
  - Research Site, Saint Petersburg
- Research Site, Singapore, Singapore
- South Korea (3):
  - Research Site, Busan
  - Research Site, Gwangju
  - Research Site, Seoul
- Spain (6):
  - Research Site, Barcelona
  - Research Site, Girona
  - Research Site, Madrid
  - Research Site, Marbella
  - Research Site, Santiago de Compostela
  - Research Site, Valencia
- Research Site, Lausanne, Switzerland
- Taiwan (4):
  - Research Site, Taichung
  - Research Site, Tainan
  - Research Site, Taipei
  - Research Site, Taoyuan District
- Thailand (3):
  - Research Site, Bangkok
  - Research Site, Chiang Mai
  - Research Site, Hat Yai
- Turkey (Türkiye) (4):
  - Research Site, Ankara
  - Research Site, Bursa
  - Research Site, Istanbul
  - Research Site, Izmir
- Ukraine (6):
  - Research Site, Chernivtsi
  - Research Site, Dnipro
  - Research Site, Ivano-Frankivsk
  - Research Site, Kyiv
  - Research Site, Uzhhorod
  - Research Site, Vinnytsia
- United Kingdom (2):
  - Research Site, London
  - Research Site, Sheffield
- Vietnam (3):
  - Research Site, Hanoi
  - Research Site, Ho Chi Minh City
  - Research Site, Hồ Chí Minh

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home